CLINICAL TRIAL: NCT05075083
Title: Immunogenicity and Safety of an Inactivated COVID-19 Vaccine in Elderly People With Chronic Bronchitis and Chronic Obstructive Pulmonary Disease
Brief Title: Immunogenicity and Safety of an Inactivated COVID-19 Vaccine in Elderly People With Chronic Bronchitis and COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Zhejiang Provincial Center for Disease Control and Prevention (Other Government); Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BIBP2021COPD
Record Dates: First submitted 2021-10-04; First posted 2021-10-12 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Chronic Bronchitis; COPD
MeSH Terms: conditions — COVID-19; Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: subjects aged ≥60 with chronic bronchitis and COPD receive two doses inactivated COVID-19 vaccine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): A total 400 subjects receive two doses inactivated COVID-19 vaccine with the interval of 21 days
  Interventions: Biological: Inactivated COVID-19 vaccine

INTERVENTIONS:
Biological: Inactivated COVID-19 vaccine — receive two doses inactivated COVID-19 vaccine with the interval of 21 days

SUMMARY:
Evaluation of immunogenicity and safety of the subjects aged 60 years and above with chronic bronchitis and chronic obstructive pulmonary disease recruited to receive the schedule of two doses inactivated COVID-19 vaccine with the interval of 21 days .

DETAILED DESCRIPTION:
The subjects aged 60 years and above with chronic bronchitis and chronic obstructive pulmonary disease were recruited to receive the schedule of two doses inactivated COVID-19 vaccine with the interval of 21 days .

Blood samples will be collected 2 times: before the 1st dose of vaccinatioin and 28 days after the 2nd dose of vaccination.

Any local or systemic adverse events that occurred within 21 days after vaccination will be recorded.

ELIGIBILITY:
Inclusion criteria:

* Subjects aged 60 and above with full capacity for civil conduct;
* Chronic bronchitis (or chronic obstructive pulmonary disease) diagnosed by a medical institution at level I or above;
* Body temperature < 37.3 ° C confirmed by clinical examination before enrollment ;
* Able and willing to complete the entire study plan during the study follow-up period;
* Have the ability to understand the study procedures, voluntarily sign informed consent, and comply with the requirements of the clinical study protocol

Exclusion criteria for the first dose:

* Subjects were previously confirmed cases of COVID-19 or asymptomatic infected persons;
* Subjects have history of vaccination against COVID-19;
* Being allergic to any component of vaccines (including excipients) ;
* Injection of non-specific immunoglobulin within 1 month before enrollment;
* Injection of live attenuated vaccines within 1 month and injection of other vaccines within 14 days before enrollment;
* Subjects who have experienced severe allergic reactions to vaccines (e.g. acute anaphylaxis, urticaria, angioneurotic edema, dyspnea, etc.);
* Having uncontrolled epilepsy and other progressive neurological disorders and a history of Guillain-Barre syndrome;
* Having severe liver and kidney diseases, malignant tumors, acute diseases or acute episodes of chronic diseases;
* Have been diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukaemia or other autoimmune diseases;
* Have been diagnosed with thrombocytopenia or other clotting disorders that may contraindicate subcutaneous injection;
* During an acute episode of chronic bronchitis/chronic obstructive pulmonary disease;
* Other subjects whose physical conditions, as determined by the investigator, are not suitable for inclusion in clinical studies.

Exclusion criteria for the second dose:

* Subjects who had vaccine-related adverse reactions after the first dose;
* Having high fever (axillary temperature ≥39.0℃) for three days after the first dose of inoculation, or severe allergic reaction;
* Having any adverse nervous system reaction after the first dose;
* During the acute onset of a chronic disease, or the recovery of acute complications less than two weeks;
* Other reasons for exclusion considered by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate | 28 days after the 2th dose (Day 49)
  The rate of seroconversion against coronavirus
Baseline neutralizing antibody level | Before vaccination (Day 0)
  Neutralizing antibody geometric mean titer(GMT) against coronavirus before vaccination
Neutralizing antibody level | 28 days after the 2th dose (Day 49)
  Neutralizing antibody GMT against coronavirus after the 2th dose

SECONDARY OUTCOMES:
Adverse events rate | 0-21days following vaccinations
  Analyse the incidence of adverse events following vaccination, both solicited and unsolicited
Serious adverse event rate | 0-6 months
  Report and analyse serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hanqing He, Principal Investigator — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Zhejiang provincial center for disease control and prevention, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No